CLINICAL TRIAL: NCT06821542
Title: A Phase 3, Randomized, Open-Label Study of Axatilimab Versus Best Available Therapy in Participants With Chronic Graft Versus Host Disease After at Least 2 Prior Lines of Systemic Therapy
Brief Title: A Study to Evaluate Axatilimab Versus Best Available Therapy in Participants With Chronic Graft Versus Host Disease After at Least 2 Prior Lines of Systemic Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCA034176-355; 2024-518973-32-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab; Calcineurin Inhibitors; Cyclosporine; Tacrolimus; Photopheresis; Mycophenolic Acid; Everolimus; Sirolimus; Rituximab; Pentostatin; Proteasome Inhibitors; Imatinib Mesylate; ibrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Axatilimab (Experimental): Axatilimab at the protocol-defined dose.
  Interventions: Drug: INCA034176
- Best available Treatment (BAT) (Experimental): Best Available Therapy (BAT) will be selected by the Investigator for each participant. BAT may not include experimental agents (i.e. those not approved for the treatment of any indication) as well as a limited number of other selected drugs in accordance with the protocol-defined requirements.
  Interventions: Drug: Best Available Therapy (BAT)

INTERVENTIONS:
Drug: INCA034176 — IV infusion
  Other Names: Axatilimab
  Arms: Axatilimab
Drug: Best Available Therapy (BAT) — Best Available Therapy (BAT) will be selected by the Investigator for each participant. BAT may not include experimental agents (i.e. those not approved for the treatment of any indication) as well as a limited number of other selected drugs in accordance with the protocol-defined requirements.
  Other Names: BAT could include:; • Calcineurin inhibitor (cyclosporine or tacrolimus); • Extracorporeal photopheresis (ECP); • Mycophenolate mofetil (MMF); • A mammalian target of rapamycin (mTOR) inhibitor (everolimus or sirolimus); • Rituximab; • Pentostatin; • Proteasome inhibitors; • Imatinib; • Ibrutinib
  Arms: Best available Treatment (BAT)

SUMMARY:
This study will be conducted to compare Axatilimab Versus Best Available Therapy in Participants With Chronic Graft Versus Host Disease After at Least 2 Prior Lines of Systemic Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years at the time of signing the ICF.
* Active, moderate to severe cGVHD, requiring systemic immune suppression.
* Participants with refractory or recurrent cGVHD who have received at least 2 lines of systemic therapy, including corticosteroids and ruxolitinib.
* Concomitant use of systemic corticosteroids is allowed. Participants on systemic corticosteroids must be on a stable dose of corticosteroids for at least 2 weeks prior to C1D1. Topical and inhaled corticosteroid agents are allowed.
* Participants must accept to be treated with one of the following BAT options on C1D1: CNI (cyclosporine or tacrolimus), ECP, MMF, an mTOR inhibitor (everolimus or sirolimus), rituximab, pentostatin, proteasome inhibitors, imatinib, or ibrutinib.
* History of allo-HCT from any donor HLA type (related or unrelated donor with any degree of HLA matching) using any graft source (bone marrow, peripheral blood stem cells, or cord blood). Recipients of myeloablative, nonmyeloablative, or reduced-intensity conditioning are eligible.

Exclusion Criteria:

* Receipt of more than 1 prior allo-HCT. Prior autologous HCT is allowed.
* Evidence of relapse of hematologic disease or treatment for relapse after the allo-SCT was performed, including DLI for the treatment of molecular relapse. Note: Participants who have received a scheduled DLI as part of their transplant procedure and not for management of malignancy relapse are eligible.
* Systemic treatment with CNIs or mTOR inhibitors started within 2 weeks prior to C1D1.
* Severe renal impairment, that is, estimated creatinine clearance < 30 mL/min measured or calculated by Cockcroft-Gault equation in adults and Schwartz formula in pediatric participants, or end-stage renal disease on dialysis.
* Impaired liver function, defined as total bilirubin > 1.5 × ULN and/or ALT and AST > 3 × ULN in participants with no evidence of liver cGVHD.
* History of acute or chronic pancreatitis.
* Active, symptomatic myositis.
* Pregnant or breastfeeding.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2025-06-04 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) at 6 months | 6 months
  Defined for each treatment group as complete response (CR) or partial response (PR) at 6 months (Cycle 7 Day 1, 28-day cycles) in the absence of new systemic therapy for cGVHD. Responses defined by the 2014 NIH consensus criteria.

SECONDARY OUTCOMES:
Failure-free survival (FFS) | Up to 5 years
  Defined as the time from the date of randomization to the date of addition or initiation of another systemic therapy for cGVHD, relapse of underlying disease, or death due to any cause.
Proportion of participants with a ≥ 7-point improvement in modified Lee Symptom Scale (mLSS) total score | Up to 5 years
Overall Response at 12 months | 12 months
  Defined as CR or PR at 12 months in the absence of new systemic therapy for cGVHD.
Best Overall Response (BOR) | Up to 5 years
  Defined as the best response of CR or PR in the first 6 months (up to and including Cycle 7 Day 1), and at any timepoint up to the initiation of new therapy for cGVHD.
DOR (in responders only) | Up to 5 years
  Defined as the time from the date of first response (PR or CR) to the date of progression of cGVHD from baseline scoring, start of new systemic treatment for cGVHD, or death from any cause, whichever comes first. An additional measure of response durability will consider DOR as the time from the date of first response to the date of new systemic therapy for cGVHD or death from any cause, whichever occurs first.
Organ-specific response | Up to 5 years
  Organ-specific response as defined in the protocol.
Overall Survival (OS) | Up to 5 years
  Defined as the time from the date of randomization to the date of death due to any cause.
Nonrelapse mortality (NRM) | Up to 5 years
  Defined as the time from the date of randomization to the date of death not preceded by relapse of primary hematologic disease.
Time to primary hematologic disease relapse | Up to 5 years
  Defined as the time from the date of randomization to the date of relapse.
Percent reduction in daily corticosteroid dose at 6 months | 6 months
Proportion of participants who tapered off all corticosteroids at 6 months | 6 months
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 5 years and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after the first dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (130):
- Austria (5):
  - Medical University of Graz, Graz
  - Medizinische Universitaet Innsbruck - Universitaetsklinik Fuer Innere Medizin Iii, Innsbruck
  - Krankenhaus Der Elisabethinen Linz Gmbh, Linz
  - Medizinische Universitat Wien, Universitatsklinik Fur Innere Medizin I, Vienna
  - St. Anna Childrens Hospital, Vienna
- Belgium (6):
  - Az Sint-Jan Brugge Av, Bruges
  - Chu Ucl Namur Site Godinne, Godinne-mont
  - Universitair Ziekenhuis Leuven, Leuven
  - Chu Liege -Centre Hospitalier Universitaire Sart Tilman, Liège
  - Algemeen Ziekenhuis Delta, Roeselare
  - Universite Catholique de Louvain (Ucl) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Czechia (3):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava-poruba
  - Ustav Hematologie A Krevni Transfuze (Uhkt), the Institute of Hematology and Blood Transfusion (Ihbt, Prague
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - New Children'S Hospital, University of Helsinki and Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku
- France (14):
  - Chu D'Amiens-Picardie - Hopital Sud, Amiens
  - CHU CAEN, Caen
  - Centre Hospitalier Regional Universitaire (Chru) de Lille - Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - Chu de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice,Hopital L Archet, Nice
  - Hospital Saint-Louis - Aphp, Paris
  - Hopital Universitaire Robert Debre, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud Cancer Comprehensive Center - Iuct Oncopole, Toulouse
  - Chru Nancy, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus Grand Paris- (Institut de Cancerologie Gustave-Roussy), Villejuif
- Germany (17):
  - Uniklinik Rwth Aachen Medizinische Klinik Iv, Aachen
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - University Hospital Carl Gustav Carus, Dresden
  - Universitatsklinikum Erlangen, Erlangen
  - Klinikum Der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsmedizin Goettingen, Göttingen
  - Universitaetsklinikum Halle, Halle
  - Universitaetsklinikum Des Saarlandes, Homburg
  - Universitaetsklinikum Schleswig-Holstein, Uksh-Campus Kiel, Kiel
  - University Hospital Leipzig, Leipzig
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Universitaetsklinikum Muenster, Münster
  - University Clinic Regensburg, Regensburg
  - University Hospital of Ulm, Universitatsklinikum Ulm, Ulm
  - University of Wuerzburg, Würzburg
- Greece (4):
  - General Hospital of Athens Evangelismos - Eye Hospital, Athens
  - Attikon Hospital and Cutaneous Lymphoma Clinic-Athens University Medical School, Athens
  - University Hospital of Patras, RIO Patras
  - General Hospital of Thessalonikis George Papanikolaou - Gene and Cell Therapy Center, Thessaloniki
- St. James Hospital, Dublin, Ireland
- Italy (31):
  - Ss Antonio & Biagio and C. Arrigo Hospital, Alessandria
  - Azienda Ospedaliero Universitaria Delle Marche Clinica Ematologica, Ancona
  - Azienda Ospedaliera Papa Giovanni Xxiii, Bergamo
  - Azienda Ospedaliera Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S. Orsola-Malpighi - Istituto Di Ematolog, Bologna
  - Universita Degli Studi Di Brescia - Azienda Ospedaliera Spedali Civili Di Brescia, Brescia
  - Azienda Policlinico Vittorio Emanuele, Presidio G Rodolico, Universita Di Catania, Catania
  - Azienda Ospedaliero Universitaria Careggi-S.O.D. Patologia Medica, Florence
  - Irccs - Azienda Ospedaliera Universitaria - Ist San Martino, Genova
  - Pia Fondazione Cardinale Giovanni Panico Azienda Ospedaliera, Lecce
  - Fondazione Irccs Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) - Ospedale San Raffaele (Hsr) (Istituto, Milan
  - Asst Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera San Gerardo Di Monza, Monza
  - Azienda Ospedaliero Universitaria Federico Ii Di Napoli, Naples
  - Azienda Ospedaliera Di Rilievo Nazionale (Aorn) 'Antonio Cardarelli', Napoli
  - Azienda Ospedale Universita Di Padova, Padua
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Irccs Fondazione Policlinico San Matteo, Pavia
  - Presidio Ospedaliero Spirito Santo Azienda U.S.L. Pescara, Pescara
  - Morelli Hospital, Reggio Calabria
  - Aou Policlinico Umberto I, Roma
  - A. Gemelli University Hospital, Catholic University of the Sacred Heart, Roma
  - Fondazione Ptv Policlinico Tor Vergata, Rome
  - Irccs Ospedale Pediatrico Bambino Gesu, Rome
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Fondazione Ircss Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - A.O.U. Citta Della Salute E Della Scienza Di Torino, Torino
  - Ospedale Santa Maria Di Ca' Foncello, Treviso
  - Clinica Ematologica, Dism Azienda Ospedaliero Universitaria, Udine
  - Uoc Ematologia E Centro Trapianti Midollo Osseo Br, Ospedale Borgo Roma, Verona
- Netherlands (6):
  - Amsterdam University Medical Center (Amsterdam Umc), Vrije University Medical Center (Vumc), Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center (Leids Universitair Medisch Centrum (Lumc)), Leiden
  - Maastricht University Medical Center (Mumc), Maastricht
  - Erasmus Medisch Centrum 1, Rotterdam
  - Universitair Medisch Centrum Utrecht (Umc Utrecht), Utrecht
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Rikshospitalet University Hospital, Oslo
- Portugal (3):
  - Ipo Lisboa Francisco Gentil, Lisbon
  - Centro Hospitalar Universitario Lisboa Norte Epe, Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil E.P.E, Porto
- Spain (21):
  - Institut Catala D'Oncologia Badalona, Hospital Germans Trias I Pujol, Badalona
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona (Hospital Clinic I Provincial), Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Institut Catala D Oncologia, Barcelona
  - Hospital Clinico Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Sant Joan de Deu Barcelona - Children'S Hospital, Esplugues de Llobregat
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Maranon (Hgugm), Madrid
  - Hospital Universitario Infantil Nino Jesus, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario de Donostia, SAN Sebasttian
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario de Valencia (Instituto de Investigacion Sanitaria Incliva), Valencia
  - Universitat de Valencia - Hospital Universitari I Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - University of Gothenburg and Queen Silvia Children S Hospital At Sahlgrenska University Hospital, Gothenburg
  - Skanes Universitetssjukhus - Universitetssjukhuset I Lund, Lund
  - Karolinska Universitetssjukhuset, Centrum For Cellterapi Och Allogen Stamcellstransplantation, Stockholm
  - Uppsala University Hospital, Uppsala
- Switzerland (4):
  - University Hospital Basel, Basel
  - Hopitaux Universitaires de Geneve (Hug) - Centre de Recherche Clinique (Crc), Geneva
  - Universitatsspital Zurich, Zurich
  - Universitats-Kinderspital Zurich Eleonorenstiftung, Zurich
- United Kingdom (5):
  - Cardiff and Vale Nhs Trust - University Hospital of Wales (Uhw), Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - St James'S University Hospital - Leeds Teaching Hospitals Nhs Trust, Leeds
  - University Hospitals of Leicester Nhs Trust-Leicester Royal Infirmary, Leicester
  - King'S College Hospital Nhs Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate Axatilimab Versus Best Available Therapy in Participants With Chronic Graft Versus Host Disease After at Least 2 Prior Lines of Systemic Therapy — https://www.incyteclinicaltrials.com/study/?id=INCA034176-355&SearchTerm=INCA034176-355&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=